CLINICAL TRIAL: NCT03769428
Title: Postoperative Analgesia in Breast Cancer Surgery: Safety and Efficiency of Ultrasound Guided Erector Spinae Plane Block, a Randomized Controlled Double Blinded Trial
Brief Title: Postoperative Analgesia in Breast Cancer Surgery: Safety and Efficiency of Ultrasound Guided Erector Spinae Plane Block
Acronym: erectspinae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben marzouk Sofiene (Other)
Responsible Party: Sponsor-Investigator, Ben marzouk Sofiene, clinical associate professor, University Tunis El Manar
Organization: University Tunis El Manar (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: erector-spinae
Record Dates: First submitted 2018-11-27; First posted 2018-12-07 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer Surgery; Postoperative Analgesia
Keywords: opioid consumption; erector spinae plane block; breast surgery; analgesia; PCA morphine; Locoregional anesthesia; breast cancer surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group B:ESP block (Active Comparator): Patients in the experimental arm will receive an erector spinae plane block prior to induction of general anesthetic :- 150 mg of Ropivacaine : 40cc of Ropivacaine (3.75mg/cc)
  * An intravenous patient controlled analgesia device will be given to the patients postoperatively
  Interventions: Procedure: erector spinae plane block
- group P: Sham ESP block (Placebo Comparator): Patients allocated to the placebo-control arm will receive a sham erector spinae plane block .they will receive a placebo injection of normal saline in a fashion almost identical to that of the ESP block:- 40 cc of normal saline will be injected
  -An intravenous patient controlled analgesia device will be given to the patients postoperatively
  Interventions: Procedure: sham erector spinae plane block

INTERVENTIONS:
Procedure: erector spinae plane block — The ESPB will be done in a sitting position using linear ultrasound probe (L10) of MySonoU6 machine. The blocks will be performed at the T4-T5 level of the spine using an in-plane approach. A linear probe will be placed 2-3 cm laterally to the spine using a sagittal approach. Three muscles will be identified superficial to the transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. Local anesthetic (LA) is injected between the erector spinae muscle and transverse process. Following confirmation of the correct position of the needle tip with administration of 0.5-1 ml of the fluid. Then 40cc of Ropivacaine (3.75mg/cc) will be injected .The distribution will be observed in both cranial and caudal directions.
  Arms: group B:ESP block
Procedure: sham erector spinae plane block — The sham ESPB will be done in a sitting position using linear ultrasound probe (L10) of MySonoU6 machine. The blocks will be performed at the T4-T5 level of the spine using an in-plane approach. A linear probe will be placed 2-3 cm laterally to the spine using a sagittal approach. Three muscles will be identified superficial to the transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. Following confirmation of the correct position of the needle tip with administration of 0.5-1 ml of the fluid a total of 40 mL of fluid will be injected next between the erector spinae muscle and transverse process. Then 40cc of normal saline will be injected.The distribution will be observed in both cranial and caudal directions.
  Arms: group P: Sham ESP block

SUMMARY:
Breast cancer surgery is one of the most common surgeries, due to the high incidence of breast cancer. Unfortunately, patients experience significant postoperative acute pain, placing them at risk for increased clinical morbidity and the development of disabling chronic pain which may rich up to 55% . The intensity of perioperative pain experienced by the patient is one of the best predictors of chronic pain.

However, postoperative analgesia in breast cancer surgery is difficult due to the extensive nature of the surgery and the complex innervation of the breast.

Several newly described regional anesthesia techniques exist to control perioperative pain, including the Paravertebral block (PVB) which has been proved to be the most effective one. The anatomic proximity of the pleura and central neuraxial system makes it a particularly challenging technique and carrying a risk of pneumothorax.

The Erector Spinae Plane Block (ESPB) is a novel interfascial plane block described by Forero et al in September 2016. Local anesthetic injection is performed beneath the erector spinae muscle. Local anesthetic (LA) expected to achieve paravertebral spread of three vertebral levels cranially and four levels caudally, blocking the dorsal and ventral rami of the spinal nerves.The easy, fast and safe execution of ESPB makes it a promising technique in the context of surgical pain during breast cancer surgery.

There is no sufficient randomized controlled trials that assess the effectiveness of ESPB in controlling post-operative breast surgery pain.

The main purpose of this study is to evaluate the postoperative analgesic effect of Ultrasound-guided ESPB in patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
It is a prospective double blind trial. Sixty female patient aged between 20-65 years old with American Society of Anesthesiologists (ASA) physical status I-II and scheduled for elective surgery for breast cancer were included in the study. Only unilateral surgical procedures will be included. The patients will be randomized into two groups:

Group B (ESP block): Patients in the experimental arm will receive an ESPB prior to induction of general anesthetic.

Group P: (sham ESP block): Patients allocated to the placebo-control arm will receive a placebo injection of normal saline in almost identical fashion to that of the ESP block.

Intravenous access will be obtained with an 18-gauge intravenous (IV) cannula in the contralateral upper limb of the surgical site and monitors (pulse oximeter, electrocardiography, non-invasive blood pressure (NIBP) will be applied.

All blocks will be performed before induction of general anesthesia.

ESPB technique:

The ESPB will be done in the sitting position using linear ultrasound probe (L10) of MySonoU6 machine. The blocks will be performed at the T4-T5 level of the spine using an in-plane approach. A linear probe will be placed 2-3 cm laterally to the spine using a sagittal approach. Three muscles will be identified superficial to the transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. Local anesthetic (LA) is injected between the erector spinae muscle and transverse process. Following confirmation of the correct position of the needle tip with administration of 0.5-1 ml of the fluid a total of 40 mL of fluid will be injected next. The distribution will be observed in both cranial and caudal directions.

* Group B (ESP block) will receive 150 mg of Ropivacaine : 40cc of Ropivacaine (3.75mg/cc).
* Group P (Sham ESP block) will receive 40 cc of normal saline.

General Anesthesia:

All patients will receive pre-oxygenation with 100% O2 for 3 min. Anesthesia will be induced by using fentanyl 2μg/kg, Propofol 2-3 mg/kg and Atracurium 0.5 mg/kg. During anesthesia maintenance, monitoring will include Pulse Oximetry, an Electrocardiogram, Non-Invasive Blood Pressure (NIBP), end-tidal Carbon Dioxide, End-Tidal Sevoflurane, and Fraction of Inspired Oxygen.

The reinjection of 0.5μg/kg of fentanyl will be given intraoperatively either when heart rate or Non-Invasive Blood Pressure (NIBP) report an increase by more than 20% of the basal records.

Paracetamol 1 g IV and Ketoprofen 100 mg intramuscular (IM) will be administered for postoperative analgesia at the end of surgery. Anesthesia will be discontinued and tracheal extubation will be done once patient fulfilled the extubation criteria. In the recovery room, all patients will be given a patient-controlled analgesia device (PCA) containing morphine 1 mg/ml-1 ,set to deliver a 1 mg bolus dose of morphine, with an 5 min lockout time and 12mg 1 h limit. Postoperative pain will be assessed using a visual analogue scales (VAS) scores ranging from zero (no pain) to 10 (worst imaginable pain). The VAS scores will be recorded at 1,2,4,8 6, 12, 16, 20 and 24 h postoperatively.If VAS scores are superior to 6 the investigators will resort to rescue analgesia as following: If 6<VAS<8: paracetamol 1g IV will be administered and if VAS>8: paracetamol 1g IV associated to ketoprofen100mg IM.

Incidence of nausea and vomiting, and total morphine consumption during the 24-h postoperative period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old
* ASA I-II
* Undergoing unilateral breast cancer surgery

Exclusion Criteria:

* obesity (body mass index >40 kg/m2)
* Preoperative chronic dependence upon opioid and NSAID medications
* History of psychiatric or neurological disease
* Patients with chronic pain syndromes
* allergy to local anaesthetics
* other contraindications to peripheral nerve blocks
* Patients' refusal to participate

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Comparing morphine consumption rates within 24h postoperative | The first 24 hours postoperative
  All patients will be provided with IV morphine PCA and morphine consumption within 24 hour postoperatively will be recorded for both groups.

SECONDARY OUTCOMES:
Assessment of pain in postoperative period via visual analogue scales (VAS) . | The first 24 hours postoperative
  Postoperative pain will be assessed using a VAS ranging from 0 (no pain) to 10 (worst imaginable pain).The VAS will be recorded at 1,2,4,8 6, 12 ,16,20 and 24 h postoperatively.
Total morphine demand | During 24 hours postoperative
  The investigators will compare total morphine demand in both groups during the first 24h after surgery.
Time to first request for morphine | During 24 hours postoperative
  The investigators will compare the timing of the first request for morphine in both groups during the first 24h after surgery.
Requirement of rescue analgesia | During 24 hours postoperative
  The investigators will record and compare the timing of first rescue analgesia and total rescue analgesia requirement.
  If 6<VAS<8: paracetamol 1g iv will be administered If VAS>8:paracetamol 1g iv associated to ketoprofen100mg IM will be administered.
Total intraoperative consumption of Fentanyl. | Intraoperative period
  The investigators will record the total dose of Fentanyl (µg) required during surgery.
  Fentanyl will be given intraoperatively either when heart rate or Non-Invasive Blood Pressure (NIBP) report an increase by more than 20% of the basal records.
Postoperative nausea and vomiting | within 24 hours postoperative
  Incidence of postoperative nausea and vomiting will be recorded.
Morphine related side effects | During 24 hours postoperative
  The occurence of morphine related side effects such as pruritus,urinary retention,hypotension,respiratory distress and sedation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hayen Maghrebi, PROFESSOR, Study Chair — UNIVERSITY OF TUNIS EL MANAR
Locations (1):
- Tunis maternity and neonatology center,, Tunis, Tunisia